CLINICAL TRIAL: NCT00933205
Title: An Open Label Safety Study of Tipranavir Co-administered With Low-dose Ritonavir (TPV/r) in Patients With Advanced HIV-1 Infection and Limited Treatment Options.
Brief Title: An Open Label Safety Study of Tipranavir Co-administered With Low-dose Ritonavir in Patients With Advanced HIV-1 Infection and Limited Treatment Options.
Status: Approved for marketing | Type: Expanded Access
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Other Study IDs: 1182.16
Record Dates: First submitted 2009-07-03; First posted 2009-07-07 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2013-10

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — tipranavir

INTERVENTIONS:
Drug: Tipranavir

SUMMARY:
The purpose of this Open Label Safety Study is to provide access to and evaluate the safety and tolerability of TPV/r in treatment-experienced patients with advanced HIV-1 infection who have failed at least two PI-containing regimens, and have limited treatment options.

ELIGIBILITY:
Inclusion Criteria:

1. Triple anti-retroviral class experienced patients with at least 2 previous PI-based regimens who had failed or are intolerant to currently approved HIV-1 treatments.
2. Age equal or more than 18 years
3. Patient is willing to use an effective barrier method of contraception for the duration of study participation and up to three months thereafter
4. Patient voluntarily provides written informed consent to participate, in compliance with local law.

Exclusion Criteria:

1. Hypersensitivity to active ingredients or any of the excipients in tipranavir or ritonavir
2. Required use of restricted medications.
3. Female patients of childbearing potential who have a positive pregnancy test at baseline or are breast feeding.
4. Any medical condition which in the opinion of the investigator would interfere with the patients' ability to participate in or adhere to the requirements of this protocol.
5. Use of other investigational drugs, within 30 days prior to TPV boosted with ritonavir initiation and for the duration of study participation
6. Hepatic impairment evidenced by the following baseline laboratory findings:

   * AST or ALT more than 5X ULN or total bilirubin more than 3.5X ULN
   * AST or ALT more 2.5X ULN and total bilirubin more 2X ULN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-05; Primary Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (215):
- Belgium (11):
  - 1182.16.3202 Boehringer Ingelheim Investigational Site, Antwerp
  - 1182.16.3203 Boehringer Ingelheim Investigational Site, Brussels
  - 1182.16.3205 Boehringer Ingelheim Investigational Site, Brussels
  - 1182.16.3206 Boehringer Ingelheim Investigational Site, Brussels
  - 1182.16.3207 Boehringer Ingelheim Investigational Site, Brussels
  - 1182.16.3211 Boehringer Ingelheim Investigational Site, Charleroi
  - 1182.16.3204 Boehringer Ingelheim Investigational Site, Ghent
  - 1182.16.3201 Boehringer Ingelheim Investigational Site, Leuven
  - 1182.16.3208 Boehringer Ingelheim Investigational Site, Liège
  - 1182.16.3212 Boehringer Ingelheim Investigational Site, Liège
  - 1182.16.3209 Boehringer Ingelheim Investigational Site, Luxembourg
- Brazil (12):
  - 1182.16.5511 Unidade de Pesquisa Clínica (UPC) - AIDS, Campinas - Sp
  - 1182.16.5505 Hospital São José de Doenças Infecciosas de Fortaleza, Fortaleza - Ce
  - 1182.16.5502 Hospital Nossa Senhora da Conceiç, Porto Alegre - Rs
  - 1182.16.5504 Hospital das Clínicas de Porto Alegre, Porto Alegre - Rs
  - 1182.16.5512 Ambulatório de DST/ AIDS - RS, Porto Alegre - Rs
  - 1182.16.5513 Centro de Pesquisa Hospital Evandro Chagras, Rio de Janeiro
  - 1182.16.5509, Rio de Janeiro - Rj
  - 1182.16.5510, Santos - Sp
  - 1182.16.5501 UNIFESP/ Hospital São Paulo- Univers. Federal de São Paulo, São Paulo - Sp
  - 1182.16.5506 Casa da AIDS da FMUSP, São Paulo - Sp
  - 1182.16.5507 Hospital do Servidor Público Estadual de São Paulo, São Paulo - Sp
  - 1182.16.5508, Vila Mariana
- Canada (26):
  - 1182.16.1118, Calgary, Alberta
  - 1182.16.1104 University of Alberta H-Site, Edmonton, Alberta
  - 1182.16.1101 St. Paul's Hospital, Vancouver, British Columbia
  - 1182.16.1111 Downtown Infectious Diseases Clinic, Vancouver, British Columbia
  - 1182.16.1125 St. Boniface General Hospital, Winnipeg, Manitoba
  - 1182.16.1131 The Moncton Hospital, Moncton, New Brunswick
  - 1182.16.1128 Centre for Clinical Research, Halifax, Nova Scotia
  - 1182.16.1112 McMaster University Medical Centre, Hamilton, Ontario
  - 1182.16.1126 HIV Care Programme, London, Ontario
  - 1182.16.1132 Infectious Diseases Consultant, Oakville, Ontario
  - 1182.16.1102 Canadian Immunodeficiency Research Collaborative Inc., Toronto, Ontario
  - 1182.16.1107 Sunnybrook & Woman's College Health Science Centre, Toronto, Ontario
  - 1182.16.1109 Infectious Diseases and HIV, Toronto, Ontario
  - 1182.16.1110 Toronto East General Hospital, Toronto, Ontario
  - 1182.16.1114 Toronto General Hospital, Toronto, Ontario
  - 1182.16.1115, Toronto, Ontario
  - 1182.16.1124, Toronto, Ontario
  - 1182.16.1106 Positive Care Clinic, Whitby, Ontario
  - 1182.16.1120 Metropolitan Campus, Windsor, Ontario
  - 1182.16.1116 Immune Deficiency Treatment Centre, Monteal, Quebec
  - 1182.16.1103 Hopital Notre Dame CHUM, Montreal, Quebec
  - 1182.16.1113 Montreal Chest Institute, McGill University Health Centre, Montreal, Quebec
  - 1182.16.1117 Clinique medicale l'Actuel, Montreal, Quebec
  - 1182.16.1119, Montreal, Quebec
  - 1182.16.1122 Infectious Diseases, Montreal, Quebec
  - 1182.16.1130 Clinique Medicale LORI, Montreal, Quebec
- Denmark (3):
  - 1182.16.4501 Boehringer Ingelheim Investigational Site, Copenhagen
  - 1182.16.4502 Boehringer Ingelheim Investigational Site, Hvidovre
  - 1182.16.4504 Boehringer Ingelheim Investigational Site, Odense C
- El Salvador (2):
  - 1182.16.3491 Boehringer Ingelheim Investigational Site, Vic (Barcelona)
  - 1182.16.3464 Boehringer Ingelheim Investigational Site, Vizcaya
- Greece (8):
  - 1182.16.3001 "Andreas Syggros"Hospital of Dermatological & Veneral Diseas, Athens
  - 1182.16.3002 "Greek Red Cross" Hospital, 3rd Internal Medicine Clinic, Athens
  - 1182.16.3004 "Attiko" Hospital, 4th Internal Medicine Clinic, UOA, Athens
  - 1182.16.3005 Laiko Hospital, 2nd District Blood Donation Center & Haemato, Athens
  - 1182.16.3007 1st Social Insurance Foundation (IKA) Pentelis, Athens
  - 1182.16.3010 University Hospital of Patras, Pátrai
  - 1182.16.3008 "Tzanio" Hospital, Piraeus
  - 1182.16.3009 AHEPA Hospital, Thessaloniki
- Italy (65):
  - 1182.16.3932 Azienda Ospedaliera Umberto I, Ancona
  - 1182.16.3923 Ospedale Santa Maria Annunziata, Antella (fi)
  - 1182.16.3952 Centro di riferimento oncologico, Aviano - PD
  - 1182.16.3958 A.O. Ospedale Clinico Consorziale, Bari
  - 1182.16.3920 Ospedali Riuniti di Bergamo, Bergamo
  - 1182.16.3946 Ospedale Policlinico S. Orsola Bologna, Bologna
  - 1182.16.3938 Ospedale Civile Regionale, Bolzano
  - 1182.16.3901 Università di Brescia, Brescia
  - 1182.16.3957 A.O. Spedali Civili di Brescia, Brescia
  - 1182.16.3928 Azienda Ospedaliera, Busto Arsizio (va)
  - 1182.16.3964 Ospedale SS. Trinità, Cagliari
  - 1182.16.3947 U.O. Malattie Infettive, Catania
  - 1182.16.3961 Ospedale Pugliese, Catanzaro
  - 1182.16.3954 Ospedale Civile, Cuggiono-MI
  - 1182.16.3963 Azienda Ospedaliera Arcispedale S. Anna, Ferrara
  - 1182.16.3924 Azienda Ospedaliera Careggi, Florence
  - 1182.16.3902 Ospedali Riuniti di Foggia, Foggia
  - 1182.16.3911 U.O. di Malattie Infettive, Foggia
  - 1182.16.3926 Azienda Ospedaliera, Genova
  - 1182.16.3927 Azienda Ospedaliera, Genova
  - 1182.16.3929 Malattie Infettive, Genova
  - 1182.16.3912 Ospedale "A. Manzoni", Lecco
  - 1182.16.3925 Azienda Ospedaliera Carlo Poma, Mantova
  - 1182.16.3951 Ospedale Civile Umberto I, Mestre-VE
  - 1182.16.3903 Ospedale L. Sacco, Milan
  - 1182.16.3904 Ospedale Luigi Sacco, Milan
  - 1182.16.3910 Ospedale Luigi Sacco, Milan
  - 1182.16.3913 Fondazione Centro S. Raffaele del Monte Tabor, Milan
  - 1182.16.3953 ospedale Niguarda, Milan
  - 1182.16.3965 Ospedale Maggiore, Milan
  - 1182.16.3968 Azienda Ospedaliera Policlinico, Modena
  - 1182.16.3934 Azienda Ospedaliera D. Cotugno, Napoli
  - 1182.16.3937 Azienda Ospedaliera D. Cotugno, Napoli
  - 1182.16.3942 Azienda Ospedaliera di Padova, Padua
  - 1182.16.3914 Presidio Ospedaliero di Verbania, Pallanza (Verbania)
  - 1182.16.3948 U.O. Malattie Infettive ed Epatologia, Parma
  - 1182.16.3909 I.R.C.C.S. Policlinico San Matteo, Pavia
  - 1182.16.3921 IRCCS Policlinico San Matteo, Pavia
  - 1182.16.3966 Policlinico Monteluce, Perugia
  - 1182.16.3955 Ospedale San Salvatore, Pesaro
  - 1182.16.3967 Ospedale Civile dello Spirito Santo, Pescara
  - 1182.16.3944 Ospedale Cisanello, Pisa
  - 1182.16.3931 Ospedale Santa Maria delle Croci, Ravenna
  - 1182.16.3930 Arcispedale S. Maria Nuova, Reggio Emilia
  - 1182.16.3905 IRCCS Lazzaro Spallanzani, Roma
  - 1182.16.3906 IRCCS Lazzaro Spallanzani, Roma
  - 1182.16.3907 IRCCS Lazzaro Spallanzani, Roma
  - 1182.16.3908 IRCCS Lazzaro Spallanzani, Roma
  - 1182.16.3915 Azienda Policlinico Umberto I, Roma
  - 1182.16.3922 Università "La Sapienza", Roma
  - 1182.16.3941 Istituto Nazionale per le Malattie Infettive, Roma
  - 1182.16.3960 Università Cattolica del Sacro Cuore, Roma
  - 1182.16.3945 Istituto Malattie Infettive Università Di Sassari, Sassari
  - 1182.16.3970 Ospedale San Giuseppe Moscati, Statte (ta)
  - 1182.16.3917 Ospedale Amedeo di Savoia, Torino
  - 1182.16.3918 Ospedale Amedeo di Savoia, Torino
  - 1182.16.3919 Ospedale Amedeo di Savoia, Torino
  - 1182.16.3933 Azienda Ospedaliera Umberto I, Torrette Di Ancona
  - 1182.16.3939 Ospedale Regionale, Torrette Di Ancona
  - 1182.16.3940 Presidio Ospedaliero Cà Foncello, Treviso
  - 1182.16.3943 Policlinico Universitario di Udine, Udine
  - 1182.16.3916 Ospedale di Circolo e Fondazione Macchi, Varese
  - 1182.16.3950 Ospedale SS. Giovanni e Paolo, Venezia
  - 1182.16.3949 Policlinico Rossi "Borgo Roma", Verona
  - 1182.16.3959 Ospedale Civile di Vicenza - USSL 6, Vicenza
- Portugal (5):
  - 1182.16.3502 Hospital São Francisco Xavier, Lisbon
  - 1182.16.3503 Centro Hospitalar de Lisboa, Lisbon
  - 1182.16.3505 Hospital Santa Maria, Lisbon
  - 1182.16.3501 Unidade Local de Saúde de Matosinhos, Matosinhos Municipality
  - 1182.16.3504 Hospital Joaquim Urbano, Porto
- Spain (83):
  - 1182.16.3419 Boehringer Ingelheim Investigational Site, A Coruña
  - 1182.16.3412 Boehringer Ingelheim Investigational Site, Alcalá de Henares (Madrid)
  - 1182.16.3432 Boehringer Ingelheim Investigational Site, Alicante
  - 1182.16.3484 Boehringer Ingelheim Investigational Site, Almería
  - 1182.16.3487 Boehringer Ingelheim Investigational Site, Arrecife (Lanzarote)
  - 1182.16.3474 Boehringer Ingelheim Investigational Site, Aviles (Asturias)
  - 1182.16.3440, Badalona
  - 1182.16.3454 Boehringer Ingelheim Investigational Site, Baracaldo (Vizcaya)
  - 1182.16.3438 Boehringer Ingelheim Investigational Site, Barcelona
  - 1182.16.3442 Boehringer Ingelheim Investigational Site, Barcelona
  - 1182.16.3448 Boehringer Ingelheim Investigational Site, Barcelona
  - 1182.16.3449 Boehringer Ingelheim Investigational Site, Barcelona
  - 1182.16.3463 Boehringer Ingelheim Investigational Site, Bilbao
  - 1182.16.3476 Boehringer Ingelheim Investigational Site, Cadiz
  - 1182.16.3430 Boehringer Ingelheim Investigational Site, Cartagena
  - 1182.16.3462 Boehringer Ingelheim Investigational Site, Castellon
  - 1182.16.3429 Boehringer Ingelheim Investigational Site, Córdoba
  - 1182.16.3453 Boehringer Ingelheim Investigational Site, Donostia / San Sebastian
  - 1182.16.3431 Boehringer Ingelheim Investigational Site, El Palmar (murcia)
  - 1182.16.3488 Boehringer Ingelheim Investigational Site, Gandia (Valencia)
  - 1182.16.3411 Boehringer Ingelheim Investigational Site, Getafe (Madrid)
  - 1182.16.3418 Boehringer Ingelheim Investigational Site, Gijón (asturias)
  - 1182.16.3443 Boehringer Ingelheim Investigational Site, Girona
  - 1182.16.3427 Boehringer Ingelheim Investigational Site, Granada
  - 1182.16.3428 Boehringer Ingelheim Investigational Site, Granada
  - 1182.16.3439 Boehringer Ingelheim Investigational Site, Granollers (Barcelona)
  - 1182.16.3477 Boehringer Ingelheim Investigational Site, Hospitalet de Llobregat (Barcelona)
  - 1182.16.3480 Boehringer Ingelheim Investigational Site, Huelva
  - 1182.16.3498 Boehringer Ingelheim Investigational Site, Ibiza Town
  - 1182.16.3479 Boehringer Ingelheim Investigational Site, Jaén
  - 1182.16.3423 Boehringer Ingelheim Investigational Site, Jerez de la Frontera
  - 1182.16.3445 Boehringer Ingelheim Investigational Site, L'Hospitalet de Llobregat
  - 1182.16.3436 Boehringer Ingelheim Investigational Site, La Laguna (santa Cruz de Tenerife)
  - 1182.16.3434 Boehringer Ingelheim Investigational Site, Las Palmas de Gran Canaria
  - 1182.16.3437 Boehringer Ingelheim Investigational Site, Las Palmas de Gran Canarias
  - 1182.16.3470 Boehringer Ingelheim Investigational Site, Leganés (Madrid)
  - 1182.16.3441 Boehringer Ingelheim Investigational Site, Lleida
  - 1182.16.3490 Boehringer Ingelheim Investigational Site, Logroño
  - 1182.16.3401 Boehringer Ingelheim Investigational Site, Madrid
  - 1182.16.3402 Boehringer Ingelheim Investigational Site, Madrid
  - 1182.16.3404 Boehringer Ingelheim Investigational Site, Madrid
  - 1182.16.3405 Boehringer Ingelheim Investigational Site, Madrid
  - 1182.16.3406 Boehringer Ingelheim Investigational Site, Madrid
  - 1182.16.3407 Boehringer Ingelheim Investigational Site, Madrid
  - 1182.16.3408 Boehringer Ingelheim Investigational Site, Madrid
  - 1182.16.3409 Boehringer Ingelheim Investigational Site, Madrid
  - 1182.16.3413 Boehringer Ingelheim Investigational Site, Madrid
  - 1182.16.3494 Boehringer Ingelheim Investigational Site, Manresa (Barcelona)
  - 1182.16.3426 Boehringer Ingelheim Investigational Site, Marbella (Málaga)
  - 1182.16.3493 Boehringer Ingelheim Investigational Site, Mataró
  - 1182.16.3492, Mataró (Barcelona)
  - 1182.16.3424 Boehringer Ingelheim Investigational Site, Málaga
  - 1182.16.3425 Boehringer Ingelheim Investigational Site, Málaga
  - 1182.16.3410 Boehringer Ingelheim Investigational Site, Móstoles (Madrid)
  - 1182.16.3489 Boehringer Ingelheim Investigational Site, Navarra
  - 1182.16.3472 Boehringer Ingelheim Investigational Site, Ourense
  - 1182.16.3417 Boehringer Ingelheim Investigational Site, Oviedo (Asturias)
  - 1182.16.3496 Boehringer Ingelheim Investigational Site, Palma de Mallorca
  - 1182.16.3450 Boehringer Ingelheim Investigational Site, Plama de Mallorca
  - 1182.16.3497 Boehringer Ingelheim Investigational Site, Reus (Tarragona)
  - 1182.16.3446 Boehringer Ingelheim Investigational Site, Sabadell (Barcelona)
  - 1182.16.3435 Boehringer Ingelheim Investigational Site, Santa Cruz de Tenerife
  - 1182.16.3455 Boehringer Ingelheim Investigational Site, Santander
  - 1182.16.3415 Boehringer Ingelheim Investigational Site, Santiago de Compostela
  - 1182.16.3420 Boehringer Ingelheim Investigational Site, Seville
  - 1182.16.3421 Boehringer Ingelheim Investigational Site, Seville
  - 1182.16.3422 Boehringer Ingelheim Investigational Site, Seville
  - 1182.16.3447 Boehringer Ingelheim Investigational Site, Tarragona
  - 1182.16.3495 Boehringer Ingelheim Investigational Site, Tarragona
  - 1182.16.3444 Boehringer Ingelheim Investigational Site, Terrassa
  - 1182.16.3456 Boehringer Ingelheim Investigational Site, Valencia
  - 1182.16.3457 Boehringer Ingelheim Investigational Site, Valencia
  - 1182.16.3458 Boehringer Ingelheim Investigational Site, Valencia
  - 1182.16.3460 Boehringer Ingelheim Investigational Site, Valencia
  - 1182.16.3461 Boehringer Ingelheim Investigational Site, Valencia
  - 1182.16.3403 Boehringer Ingelheim Investigational Site, Valladolid
  - 1182.16.3416 Boehringer Ingelheim Investigational Site, Vigo
  - 1182.16.3467 Boehringer Ingelheim Investigational Site, Vigo (Pontevedra)
  - 1182.16.3482 Boehringer Ingelheim Investigational Site, Villajoyosa (alicante)
  - 1182.16.3483 Boehringer Ingelheim Investigational Site, Vitoria-Gasteiz
  - 1182.16.3471 Boehringer Ingelheim Investigational Site, Zamora
  - 1182.16.3451 Boehringer Ingelheim Investigational Site, Zaragoza
  - 1182.16.3452 Boehringer Ingelheim Investigational Site, Zaragoza